CLINICAL TRIAL: NCT05628792
Title: In Vivo Depiction Of Bone Vascularization With UHR-CT CT And Deep Learning Algorithm Reconstruction: A Preliminary Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GILLET Romain, MD, MSK Radiologist, Central Hospital, Nancy, France
Other Study IDs: N°2-RCB/EUDRACT
Record Dates: First submitted 2022-10-28; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Bone Vascular Tumor
Keywords: CT; Osteoid Osteoma; Ultra High Resolution CT
MeSH Terms: conditions — Osteoma, Osteoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT — Ultra High Resolution CT scan

SUMMARY:
To evaluate the image quality and ability to depict in vivo bone vascularization with an ultra-high-resolution computed tomography (UHR-CT) scanner using a deep learning reconstruction (DLR) and hybrid iterative reconstruction (HIR) algorithms, compared to simulated conventional CT, using osteoid osteoma (OO) as a model.

ELIGIBILITY:
Inclusion Criteria:

* Proven osteoid osteoma
* Ultra High Resolution CT

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective inclusion of all histologically proven Osteoid Osteoma referred to our department for CT imaging
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of cortical vessels | Retrospective review of all ultra high resolution CT of the precedent 2 years
  Number
Number of nidus vessels | Retrospective review of all ultra high resolution CT of the precedent 2 years
  Number

SECONDARY OUTCOMES:
Confidence Score | Retrospective review of all ultra high resolution CT of the precedent 2 years
  1 (weak) to 5 (strong)

IPD SHARING:
Plan to Share IPD: No